CLINICAL TRIAL: NCT00001475
Title: A Randomized Trial of Interleukin-2 With or Without a Tumor Necrosis Factor Antagonist in Patients With HIV-1 Infection
Brief Title: Home Treatment of HIV-Infected Patients With Interleukin-2 With or Without a Tumor Necrosis Factor Antagonist
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 950133; 95-I-0133
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-06

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infection
Keywords: AIDS; Cytokines; Thalidomide; Monoclonal Antibody; Immunomodulator
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Interleukin-2; Thalidomide

INTERVENTIONS:
Drug: IL-2 plus Anti-TNF or Thalidomide

SUMMARY:
Patients enrolled in NIH protocol 95-I-0133 at the Clinical Center may participate in an extension phase of this study in which the drug prednisone will be eliminated from the treatment regimen. Prednisone is associated with avascular necrosis, a condition that has been found in a number of patients in this study. Also, certain patients in this protocol may receive future interleukin-2 treatment cycles at home. Home administration of IL-2 injections involves less frequent data and safety monitoring and no medical evaluations at the Clinical Center except at the beginning of each cycle.

To be eligible for home administration of IL-2, patients must:

* Be enrolled in a current NIAID protocol for IL-2 therapy and have received at least 1 year of treatment on the protocol, with at least two well-tolerated outpatient cycles at a stable dose.
* Have a history of tolerable side effects while receiving IL-2 without frequent medical interventions, intravenous fluid replacement or dose reductions.
* Not have had any significant clinical or laboratory abnormalities during days 0 to 5 of the last two outpatient cycles.
* Have a strong relationship with a private physician or health-care provider who has been involved in the patient's care and is willing to help supervise the patient's care during each home IL-2 cycle.
* Live in a home with easy telephone access and have proved reliable in responding to telephone calls from clinic staff.
* Give the clinic staff contact information for a close friend or relative who will agree to serve as a caregiver during each home cycle, providing the patient non-medical assistance and checking on his or her condition daily.
* Have reasonable access to emergency medical services and a nearby medical facility.
* Have proved reliable and consistent in using sterile technique, reconstituting IL-2 vials and administering subcutaneous IL-2 injections.
* Be receiving outpatient IL-2 injections cycles at least once every 6 months as part of their normal protocol participation.
* Have access to a home weight scale and be able to weigh themselves each day for safety monitoring.

Participants will receive IL-2 cycles on the same schedule they followed in their original protocol participation. They will be seen at the Clinical Center at regularly scheduled follow-up visits between cycles and for a medical evaluation and blood drawing before the start of each cycle to determine the safety of administering the cycle. During the home cycle, the patient's case manager or other team member will place monitoring telephone calls on days 2 and 4 of the cycle and again a week later. The timing and number of these calls may change depending on the findings of ongoing assessments of their usefulness. Patients will be required to notify the study team promptly of any complications or other problems that develop with therapy.

DETAILED DESCRIPTION:
In the initial phase of this study, HIV-infected patients with CD4 counts between 200 and 500 were randomized to receive either IL-2 alone by continuous IV infusion for 5 days every 8 weeks, IL-2 plus anti-TNF antibody, or IL-2 plus thalidomide. The primary endpoints of this study are safety and tolerability of the IL-2/TNF inhibitor combination. Secondary endpoints will include changes in CD4 counts, frequency and severity of IL-2 related side effects, changes in serum TNF levels, and plasma viral load changes. The study period is one year, with an optional extension period to follow. Enrollment was for up to forty-five IL-2-naive patients.

In the amended phase of this study, up to 60 patients with HIV infection and CD4 counts equal to or greater than 350 will be studied to determine the ability of prednisone to ameliorate IL-2 related toxicity. Patients will be randomized to one of four groups: IL-2 alone; IL-2 plus prednisone; prednisone alone; no treatment. All four groups will be treated with a combination regimen of antiretrovirals to include at least one protease inhibitor. IL-2 will be dosed SQ at a starting dosage of 7.5 mlU bid x 5 days every 8 weeks, and prednisone (or placebo) will be dosed at 0.5 mg/kg/day during IL-2 cycles. Primary endpoints are frequency of IL-2 associated fatigue and fever, CD4 count changes, and viral load changes. Secondary endpoints include frequency of other IL-2 side effects, concomitant medication use, steroid associated side effects, cytokine changes during IL-2, and IL-2 total exposure in the IL-2 plus steroid vs. IL-2 plus placebo arms. The study period is one year with an optional extension period to follow.

ELIGIBILITY:
IL-2 NAIVE PATIENTS:

Documented HIV-1 infection (ELISA and Western blot positive).

18 years or older.

CD4 count greater than or equal to 200 cells per mm(3) and less than or equal to 500 cells/mm(3)

Clinical laboratory values Grade 0 or 1.

No therapy with corticosteroids, chemotherapy, pentoxifylline, thalidomide, or experimental therapy in the prior 4 weeks.

Negative urine pregnancy test within 2 weeks prior to study entry (for women of childbearing potential).

Current treatment with a stable regimen or licensed anti-retroviral therapy for at least 2 weeks.

Adequate venous access in the upper extremities for repeated blood drawing and intravenous catheter placement.

No prior IL-2 therapy.

No malignancy other than Kaposi's sarcoma. Patients with Kaposi's sarcoma are eligible, but most not have received systemic therapy for KS within 4 weeks prior to study entry.

No history of prior AIDS-defining opportunistic infection other than pulmonary TB or recurrent pneumonia.

No active substance abuse which may affect patient safety or compliance.

No patients exhibiting psychiatric disturbance or illness which in the assessment of the protocol team may affect patient safety or compliance.

No patients with significant cardiac, pulmonary, rheumatologic, thyroid, kidney, gastrointestinal or neurological disease that could either decrease absorption of oral therapy, prove a cardiovascular risk during the fluid shifts and stresses that occur with IL-2 therapy, or that could have an inflammatory/immune etiology and thus might be activated or worsened by IL-2.

No patients with hypertension requiring continuous anti-hypertensive therapy.

No pregnant or lactating patients.

Women of childbearing potential must agree to practice abstinence or use 2 forms of contraception simultaneously beginning 1 month prior to receiving study medication and continuing thereafter until 1 month after the last dose of study medication.

Men must agree to practice abstinence or use a condom when engaging in intercourse during the same time period.

Must be willing to comply with current NIH Clinical Center guidelines concerning appropriate notification by an individual of current or ongoing sexual partners and/or needle-sharing partners regarding his or her HIV-1 seropositivity and the risk of transmission of HIV-1 infection.

No history of hypersensitivity or intolerance to either IL-2 or thalidomide.

PRIOR IL-2 THERAPY PATIENTS:

Active participation in protocols 91-CC-0113 or 93-CC-0143.

Negative urine pregnancy test within 2 weeks prior to study entry (for women of childbearing potential).

No history of hypersensitivity or intolerance to thalidomide.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85
Dates: Start 1995-06; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Davey RT Jr, Chaitt DG, Piscitelli SC, Wells M, Kovacs JA, Walker RE, Falloon J, Polis MA, Metcalf JA, Masur H, Fyfe G, Lane HC. Subcutaneous administration of interleukin-2 in human immunodeficiency virus type 1-infected persons. J Infect Dis. 1997 Apr;175(4):781-9. doi: 10.1086/513971. PMID 9086130
- [Background] Kovacs JA, Vogel S, Albert JM, Falloon J, Davey RT Jr, Walker RE, Polis MA, Spooner K, Metcalf JA, Baseler M, Fyfe G, Lane HC. Controlled trial of interleukin-2 infusions in patients infected with the human immunodeficiency virus. N Engl J Med. 1996 Oct 31;335(18):1350-6. doi: 10.1056/NEJM199610313351803. PMID 8857018
- [Background] Andrieu JM, Lu W, Levy R. Sustained increases in CD4 cell counts in asymptomatic human immunodeficiency virus type 1-seropositive patients treated with prednisolone for 1 year. J Infect Dis. 1995 Mar;171(3):523-30. doi: 10.1093/infdis/171.3.523. PMID 7876597